CLINICAL TRIAL: NCT05231577
Title: 7.5F Versus 9.2F Flexible Ureteroscopy for the Treatment of 1-2cm Renal Calculi on Postoperative Infection:An International Multicenter Randomized Controlled Trial
Brief Title: 7.5F Versus 9.2F Flexible Ureteroscopy for the Treatment of 1-2cm Renal Calculi on Postoperative Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT(2022)
Record Dates: First submitted 2022-01-31; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Kidney Stones
Keywords: ureteroscopy; postoperative fever; renal calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Patients in Group 0 undergo 7.5fr ultra-fine ureteroscopy (Experimental)
  Interventions: Procedure: 7.5fr ultra-fine ureteroscopy
- Experimental: Patients in Group 2 undergo 9.2fr ureteroscopy (Experimental)
  Interventions: Procedure: 9.2fr Ureteroscopy

INTERVENTIONS:
Procedure: 7.5fr ultra-fine ureteroscopy — The patient placed the lithotomy position, placed the ureteroscope to explore the affected ureter, retrogradely placed the guide wire, and placed the 12 / 14fr ureteral sheath under X-ray monitoring until the affected ureter was close to the outlet of the renal pelvis. Group 1 patients used 7.5fr ultra-fine ureteroscopy
  Arms: Experimental: Patients in Group 0 undergo 7.5fr ultra-fine ureteroscopy
Procedure: 9.2fr Ureteroscopy — The patient placed the lithotomy position, placed the ureteroscope to explore the affected ureter, retrogradely placed the guide wire, and placed the 12 / 14fr ureteral sheath under X-ray monitoring until the affected ureter was close to the outlet of the renal pelvis. Group 2 patients used 9.2fr Ureteroscopy
  Arms: Experimental: Patients in Group 2 undergo 9.2fr ureteroscopy

SUMMARY:
Ureteroscopic lithotripsy (RIRS) is the first-line treatment for 1-2 cm upper urinary tract stones, and the stone clearance rate can reach 81.4% - 92.5%. Fever after RIRS is the most common infection after RIRS, and its incidence is up to 20%. The incidence rate of systemic inflammatory response syndrome is 6.5% - 10.3%, sepsis 0.1% - 4.3%, with the infection progressed. If there is no timely and effective intervention in the early stage of urogenic sepsis, it can progress to septic shock, and the mortality can be as high as 30% - 40%. High intrarenal pressure is an important risk factor for postoperative infection. American Urological Association (AUA) guidelines point out that controlling intrarenal pressure at an appropriate level is particularly important to prevent postoperative infection.

The use of ureteroscopic sheath in ureteroscopic surgery can effectively reduce the intrarenal pressure, which is an important measure to reduce the incidence of postoperative infection. Theoretically, the larger the space, the better the reflux effect and the lower the incidence of postoperative infection. The study showed that the incidence of ureteral sheath infection was significantly lower than that of ureteral sheath infection after operation. When using the same caliber ureteroscopic sheath, use a smaller caliber ureteroscopy to increase the space between the ureteroscopy and the ureteral sheath, promote reflux, reduce intrarenal pressure and reduce the incidence of postoperative infection. However, there is still a lack of relevant research on the effect of different caliber ureteroscopy in the treatment of renal calculi on postoperative infection.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to receive ureteroscopy
2. Aged 18-70 years. 3.1-2cm kidney stones

Exclusion Criteria:

1. Combined with middle and lower ureteral calculi, surgical operation other than RIRS is required;
2. Patients with abnormal anatomical structure, ureteral stenosis and urinary diversion, such as ectopic kidney, horseshoe kidney and duplicate kidney;
3. Patients who have undergone nephrostomy;
4. Severe cardiopulmonary insufficiency;
5. Pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
postoperative fever | ≤ 1month postoperatively
  Postoperative fever was defined as armpit temperature ≥38C

SECONDARY OUTCOMES:
Stone free rate (SFR) | 1 month after removing the pigtail stent
  2mm Non-contrast CT is obtained for all patients at one month after removing the pigtail stent to evaluate the final SFR. Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were definded as ≤ 4mm, asymptomatic, non-obstructive and non-infectious stone particles

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, Ph.D & MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong,China, China

REFERENCES:
- [Background] Elashry OM, Elbahnasy AM, Rao GS, Nakada SY, Clayman RV. Flexible ureteroscopy: Washington University experience with the 9.3F and 7.5F flexible ureteroscopes. J Urol. 1997 Jun;157(6):2074-80. doi: 10.1016/s0022-5347(01)64677-9. PMID 9146583
- [Derived] Zhong W, Zhu W, Zhao Z, Liao B, Mai H, Liu C, Wang K, Zhang X, Xu C, Zeng G. 7.5F Mini Flexible Ureteroscope in Retrograde Intrarenal Surgery: Initial Results from a Multicenter Randomized Clinical Trial. J Endourol. 2024 May;38(5):421-425. doi: 10.1089/end.2023.0540. Epub 2024 Apr 4. PMID 38299514